CLINICAL TRIAL: NCT04772638
Title: PLAY 2 - Preschoolers Learning and Active in PLAY (PLAY Extension)
Brief Title: Preschoolers Learning and Active in PLAY (PLAY Extension)
Acronym: PLAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Pooja Tandon, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00000628
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Activity, Motor
Keywords: children; physical activity; early childhood education
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster RCT with a waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLAY intervention (Experimental): The PLAY intervention with educators, parents and children
  Interventions: Behavioral: PLAY
- Wait list control (Placebo Comparator)
  Interventions: Other: Wait list control

INTERVENTIONS:
Behavioral: PLAY — This intervention focuses on promoting physical activity in preschoolers and the adults (parents and teachers) in their lives. It consists of 1) Teacher training 2) Activity trackers for children, teachers and parents and 3) text messaging with content and individualized goal setting.
  Arms: PLAY intervention
Other: Wait list control — not an active intervention
  Arms: Wait list control

SUMMARY:
The PLAY 2 Study is the continuation of an R21 pilot PLAY study. In the R21, we tested the acceptability, feasibility and initial efficacy of three early childhood education setting- based, multi-level interventions to promote preschoolers' physical activity using wearable technology and additional behavior change techniques to engage educators and parents. We have selected one of these 3 as the main intervention for the R33 portion of the grant. The intervention will contain components of teacher wellness, parent engagement, and activity level monitoring.

DETAILED DESCRIPTION:
Physical activity in early childhood is important for numerous aspects of children's health and development. Preschoolers are thought to be very active but previous studies have shown that they are sedentary for the majority of time and not getting adequate opportunities to engage in active play. Experts have recommended strategies to promote physical activity in early learning settings and to involve parents in efforts to promote active living from a young age. Through early learning settings, we may be able to change behaviors in large groups of children and particularly benefit more vulnerable children who have fewer opportunities for outdoor play and physical activity at home or in their neighborhoods. However, meaningful engagement from families is also important and research suggests that there is gap in communication and perhaps alignment between educators and parents on the topic of preschoolers' physical activity. This research uses wearable technology to monitor physical activity in children, motivate parents and educators to help create active play opportunities, and create a platform for communication and shared accountability about this important health behavior. We will focus particularly on children from lower income backgrounds who suffer from disparities in both health and educational outcomes. Our primary outcome of interest is accelerometer measured physical activity. We will also explore how changes in preschooler's physical activity relate to behavioral indicators, which are topics of great significance to early childhood educators, policy makers and parents.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-5 who attend participating preschools and their parents s are eligible.
* Teachers and staff who work at participating preschools are eligible.

Participating preschools:

1. child care centers that offer full day child care
2. at least 1 classroom for children ages 3-5

Exclusion Criteria:

- family based child care homes

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Post-intervention physical activity | 6 Month after baseline assessment
  Accelerometer measured

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Tandon, MD MPH, Principal Investigator — Seattle Childrens
Locations (1):
- Seattle Childrens, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No